CLINICAL TRIAL: NCT02964845
Title: Availability is Not Access:Recently Incarcerated Women, HIV Risk, and Substance Use Disorders
Brief Title: Women's Initiative Supporting Health Increasing Healthcare Access
Acronym: WISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Diane Morse, Associate Professor of Psychiatry and Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RSRB#63032; 1R34DA041240-01A1 (NIH)
Record Dates: First submitted 2016-10-31; First posted 2016-11-16 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WISH with CHW and referral to HFM (Experimental): Subjects will be assigned a CHW for intervention sessions along with receiving primary care from Highland Family Medicine. CHWs will use the SDT-based, trauma-specific motivational approach in the intervention to engage women during 6 sessions. The duration of the intervention is 3 months. Each session will last 1 hour and will take place in a community location. CHW's will also help facilitate primary care by linking subjects to primary care and will use electronic records to update and receive input from medical providers, and support treatment recommendations from Trillium Health. CHWs will empower women to convey their needs to providers for HIV risk reduction, SUD, co-morbidity (MH, IPV) treatment and will support autonomy and competence for treatment in the intervention sessions.
  Interventions: Behavioral: WISH with CHW and referral to HFM
- Enhanced Treatment as Usual control (Other): eTAU participants will be given an HIV risk reduction information sheet made in cooperation with Trillium Health, HIV health providers. The sheet will include sex and drug behavioral risk reduction strategies and information on obtaining PrEP. The eTAU group is also facilitated to receive healthcare by having a cell phone, a primary care clinic which accepts patients, and bus passes.
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: WISH with CHW and referral to HFM — 6 intervention counseling sessions with a peer CHW, as well as CHW facilitated linkage to primary care and HIV risk reduction.
  Arms: WISH with CHW and referral to HFM
Other: Enhanced Treatment as Usual — Linkage to Primary care.
  Arms: Enhanced Treatment as Usual control

SUMMARY:
Women recently released (RR women) from incarceration constitute a vulnerable group characterized by high rates of untreated HIV and sexually transmitted infections (STIs), substance use disorder (SUD), mental health (MH) disorders and trauma. This interconnected syndemic requires helping RR women to overcome multiple internal and structural care barriers. This R34 builds on work conducted by the PI in a NIDA-funded K23 project, in which an intervention called Women's Initiative Supporting Health (WISH) was developed to improve RR women's engagement in HIV, Hepatitis C (HCV), and primary medical care using Self Determination Theory (SDT). The proposed R34 project, a natural extension of this prior work, will conduct a pilot randomized controlled trial (RCT) of the WISH intervention to examine feasibility, acceptability, and preliminary effectiveness.

DETAILED DESCRIPTION:
The PI identified two priority needs of RR women: (1) adequate HIV/HCV prevention counseling and services, including HIV pre-exposure prophylaxis (PrEP) medications for women at high risk, and (2) primary care as an avenue to address co-occurring SUD, MH disorders, and trauma that interfere with HIV preventive care. WISH is a gender, trauma, and culturally-specific, peer-delivered intervention designed to improve health services utilization and health behaviors. The proposed pilot RCT will examine the feasibility, acceptability and preliminary effectiveness of the WISH intervention in a community setting.

The WISH intervention is grounded in Self-Determination Theory (SDT), which shows that support for autonomy increases autonomous regulation and perceived competence which mediate engagement in healthy behaviors by overcoming internal and structural barriers. A novel and exploratory aim of the proposed study is to examine whether related biologic changes vary in association with SDT mediation measures. Serum inflammatory biomarkers interleukin (IL) -6, IL-8, C-reactive protein (CRP) and coagulation marker D-dimer variations are associated with HIV vulnerability and depression, and these biomarkers have not been studied in relation to SDT.

This study will randomize RR women to the WISH intervention or enhanced treatment-as-usual (eTAU) control. WISH peer community health workers (CHW) will conduct SDT-based individual sessions with women addressing autonomy and competence regarding linkage to HIV risk reduction treatment, SUD treatment, primary care, and structural empowerment. Structurally, the peers will be a part of the primary care medical team to: (1) inform providers regarding women's treatment needs and readiness; (2) navigate RR women to link with HIV risk reduction services including prophylaxis providers; and (3) help women overcome systemic barriers to care. The investigator will examine SDT mediation measures, associated internal and structural barriers, treatment engagement and adherence, HIV risk behaviors, and inflammation. Specific aims are as follows:

Aim 1: Evaluate the feasibility and acceptability of the WISH intervention in a community setting:

Aim 1 Outcomes: Participant mixed method feedback for all study and intervention procedures.

Aim 2: Assess the preliminary effectiveness of WISH to improve engagement in and adherence to needed treatments and associated outcomes

1. Linkage to HIV prevention services; HIV risk behaviors: Assess WISH intervention effects on HIV prevention services engagement as primary outcome, adherence, and reductions in HIV risk behaviors 2a. Hypothesis: WISH intervention will show preliminary effectiveness to improve use of preventative services, including pre-exposure prophylaxis, self-reported HIV risk behaviors, and STIs
2. SUD and other tx: Examine engagement and adherence for treatment as secondary WISH outcome. Hypothesis: WISH intervention will show preliminary effectiveness to increase SUD, primary care, and MH treatment initiation, engagement, and continuity of care, and reduced substance use & MH symptoms.

Aim 3: Assess WISH mechanisms of action: Assess preliminary effect differences in known SDT mediators in relation to Aim 2 outcomes. Hypothesis: SDT measures will mediate relationship between the intervention and Aim 2 outcomes.

Exploratory Aim: Explore inflammatory biomarker outcomes of WISH: Measure serum IL-6, IL-8, CRP, and D-dimer and associated SDT mediators in intervention and control subjects. Hypotheses: IL-6, IL-8, CRP, and D-dimer levels and associated SDT mediators will correlate.

Implications: RR women are at high risk for syndemic risk factors of HIV/HCV, SUD, mental health disorders, and trauma. Yet, engagement in needed care in this group is exceedingly low and innovative interventions are needed to address this problem. To the investigator's knowledge, this is the first study to assess a SDT-based intervention designed to address urgently needed improvements in the provision and utilization of HIV and primary care services for RR persons. The intervention incorporates health behavior change, CHW training, peer-navigation, and targets biological and behavioral mechanisms of changes in HIV risk. It further develops community and training infrastructures which will lead to reduced disparities in HIV acquisition

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* >18 years old female by birth biologically
* Any HIV risk and SUD in the year prior (adjusting for incarceration during which they may have had fewer HIV risk behaviors and less access to drugs or alcohol)
* HIV/HCV negative
* Released from incarceration within the prior 1 year or to be released within 2 weeks
* Agree to release all medical/mental health/SUD treatment records for research access
* Agree to become a patient at Highland Family Medicine for primary care

Exclusion Criteria:

* Non-English speaking
* < 18 year old
* Not biologically female
* Score <2 on the Six-Item Screener (derived from the Mini-Mental Status Examination )
* Decline HIV/HCV assessment.
* Refusal to obtain primary medical care from Highland Family Medicine.
* The inability to speak or comprehend English with sufficient skill to give consent or understand interviewers.
* Apparent intoxication; psychotic behavior or the presence of severe illness or pain that interferes with participation as determined with exclusion criteria score < 2 on the Six-Item Screener

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Preliminary effectiveness of WISH to improve engagement in and adherence to needed treatments and associated outcomes | 3 years
  The investigator will qualitatively analyze intervention/interview sessions using Atlas.ti to organize thematic content complemented by framework analysis. This is one assessment.

SECONDARY OUTCOMES:
Explore inflammation biomarkers outcomes of WISH | 3 years
  The investigator will examine serum levels of IL-6.
Explore impact of WISH on inflammatory biomarker | 3 years
  The investigator will examine serum levels of IL-8.
Explore biomarker levels in relation to intervention. | 3 years
  The investigator will examine serum levels of D-dimer.
Explore serum levels of CRP | 3 years
  The investigator will examine serum levels of CRP.
Linkage to HIV prevention services; HIV risk behaviors | 3 years
  Success will be measured by demonstrated awareness of and willingness to participate.
Linkage to prevention program. | 3 years
  Success will also be measured by if subjects made an HIV prevention appointment.
HIV prevention behaviors | 3 years
  Adherence to HIV prevention strategies will be measured.
HIV risk behavior | 3 years
  Changes in HIV risk behavior scale scores will also be measured.

OTHER OUTCOMES:
Substance Use Disorder treatment engagement | 3 years
  The investigator will measure substance use as a behavioral and biological outcome.
Mental health treatment engagement | 3 years
  The investigator will report initiation rate, engagement rate and number of services received after initiation as a singular measure for continuity of care.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Morse, MD, Principal Investigator — University of Rochester; Amali Epa-Llop, PHD, Study Director — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No